CLINICAL TRIAL: NCT03008954
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effect of GSP3 on Body Weight in Overweight and Obese Subjects
Brief Title: Effect of GSP3 on Body Weight in Overweight and Obese Subjects
Acronym: FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Attiva-03
Record Dates: First submitted 2016-12-19; First posted 2017-01-04 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-02

CONDITIONS: Overweight; Obesity
Keywords: weight loss; body composition; glycemic control; satiety
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Cellulose; hydroxypropylcellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Microcyrstalline cellulose (Avicel): provided in 5 capsules (350 mg each), twice daily (BID) prior to lunch and dinner.
  Interventions: Dietary Supplement: Avicel (modified Cellulose)
- GSP3 (2.25g) (Experimental): GSP3: provided in 3 capsules (750 mg each), plus 2 placebo capsules (350 mg each), twice daily (BID) prior to lunch and dinner
  Interventions: Device: GSP3; Dietary Supplement: Avicel (modified Cellulose)
- GSP3 (3.75g) (Experimental): GSP3: provided in 5 capsules (750 mg each), twice daily (BID) prior to lunch and dinner
  Interventions: Device: GSP3

INTERVENTIONS:
Device: GSP3 — Each capsule of GSP3 (previously Attiva) contains 700 mg of a mixture of two food-grade materials: carboxymethylcellulose that is cross-linked with citric acid.
  Arms: GSP3 (2.25g); GSP3 (3.75g)
Dietary Supplement: Avicel (modified Cellulose) — Each capsule of Avicel contains approximately 350 mg of microcrystalline cellulose
  Arms: GSP3 (2.25g); Placebo

SUMMARY:
The FLOW (First Loss Of Weight) study is designed to assess the effects of repeated administration of GSP3, an investigational product, on body weight. It is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed-dose study. FLOW is being conducted in 5 medical centers in Italy, Czech Republic, and Denmark, and will randomize 123 overweight and obese adult males and females to receive either placebo, GSP3 (2.25g), or GSP3 (3.75g) in addition to a hypocaloric diet (-600 kcal/day) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) ≥ 27 and ≤ 35 (at least 30% overweight and 30% obese subjects)
2. Ability to follow verbal and written instructions
3. Informed Consent Form signed by the subjects

Exclusion Criteria:

1. Pregnancy or lactation
2. Absence of medically approved contraceptive methods in females of childbearing potential (e.g., hysterectomy, non-oral contraceptive medications or intrauterine device combined with a barrier method, two combined barrier methods such as diaphragm and condom or spermicide; bilateral tubal ligation and vasectomy are not acceptable contraceptive methods)
3. History of allergic reaction to carboxymethylcellulose, citric acid, modified cellulose, microcrystalline cellulose, and gelatin
4. Administration of investigational products within 1 month prior to Screening Visit
5. Night-shift workers
6. Subjects who stopped smoking within 6 months prior to Screening Visit or considering smoking cessation during the study
7. Subjects anticipating surgical intervention during the study
8. Known type 1 or type 2 diabetes
9. History of eating disorders including binge eating (except mild binge eater)
10. Weight change > 3 kg within 3 months prior to and during the Screening period
11. Supine systolic blood pressure (SBP) > 150 mm Hg and/or supine diastolic blood pressure (DBP) > 90 mm Hg
12. Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
13. History of gastroesophageal reflux disease
14. History of gastric or duodenal ulcer
15. History of gastroparesis
16. History of gastric bypass or any other gastric surgery
17. History of intragastric balloon
18. History of pancreatitis
19. History of hemorrhoids
20. History of malabsorption
21. Laxative users
22. History of hepatitis B or C
23. History of human immunodeficiency virus
24. History of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
25. Any other clinically significant disease interfering with the assessments of Attiva, according to the Investigator
26. Positive serum or urine pregnancy test(s) in females of childbearing potential
27. Plasma glucose ≥ 126 mg/dL (7.0 mmol/L)
28. Abnormal serum thyrotropin (TSH)
29. Serum triglycerides > 500 mg/dL (5.65 mmol/L)
30. Positive test for drugs in the urine
31. Any relevant biochemical abnormality interfering with the assessments of Attiva, according to the Investigator
32. Anti-obesity medications (including herbal preparations) within 1 month prior to Screening Visit
33. Systemic corticosteroids within 1 month prior to Screening Visit
34. Thyroid hormones or preparations within 1 month prior to Screening Visit (except in subjects on stable dose of replacement therapy for at least 1 month)
35. Any other medication known to cause weight loss or weight gain within 1 month prior to Screening Visit
36. Medications treating hypertension within 1 month prior to Screening Visit
37. Medications treating dyslipidemia within 1 month prior to Screening Visit
38. Anticipated requirement for use of prohibited concomitant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Measured at weeks 0,1,2,4,6,8,10,12,13, and follow up (week 14)
  Change from baseline in kilograms and percent (%) weight

SECONDARY OUTCOMES:
Body weight responders | 12 weeks
  Change from baseline in body weight of at least 5%
Change in waist circumference | Measured at weeks 0,1,2,4,6,8,10,12,13, and follow up (week 14)
  Change from baseline in waist circumference (centimeters)
Change in fat mass | Measured at weeks 0 and 13
  Change in percentage (%) of total mas from baseline in fat- and bone-free fat mass measured by dual energy X-ray absorptiometry (DEXA)
Change in bone-free fat mass | Measured at weeks 0 and 13
  Change in percentage (%) of total mas from baseline in fat- and bone-free fat mass measured by dual energy X-ray absorptiometry (DEXA)
Change in appetite (hunger, satiety, and fullness) | Measured at weeks 0,1,2,4,6,8,10,12,13, and follow up (week 14)
  Assessed by self-administered Visual Analog Scale (VAS)
Change in food intake | Measured at weeks 0 and 12
  Assessed by 24 hr dietary recall

OTHER OUTCOMES:
Change in plasma glucose | Measured at baseline and week 13
  Change from baseline in millimoles per liter (mmol/L)
Change in plasma glucose status (normal, impaired, diabetic) | Measured at weeks 0 and 13
Change in serum insulin | Measured at weeks 0 and 13
  Change from baseline in miliunits per liter (mU/L)
Change in insulin resistance | Measured at weeks 0 and 13
  Change from baseline in homeostatic model assessment of insulin resistance (HOMA-IR)
Change in glycosylated hemoglobin (HbA1c) | Measured at weeks 0 and 13
  Measured in percentage (%)
Change in total cholesterol, serum low-density lipoprotein (LDL), high-density lipoprotein (HDL), total cholesterol/HDL ratio, and triglycerides | Measured at weeks 0 and 13
  measured in mg/dL
Change vital signs: heart rate, supine and standing systolic and diastolic blood pressure (SBP, DBP) | Measured at weeks 0,1,2,4,6,8,10,12,13, and follow up (week 14)
  Measured in beats per minute (heart rate) or millimeters of mercury (mmHg) for blood pressure
All adverse events (AE), serious adverse events (SAE), and gastrointestinal symptoms | Measured at weeks 0,1,2,4,6,8,10,12,13, and follow up (week 14)
  Number and % of subjects with AE/SAEs spontaneously reported; gastrointestinal symptoms solicited via questionnaire
Change in serum sodium | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline in millimoles per liter (mmol/L)
Change in serum potassium | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in serum coloride | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in serum calcium | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in serum magnesium | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in serum phosphorus | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in serum glucose | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in blood urea nitrogen (BUN) | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (mmol/L)
Change in serum creatinine | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline in micromoles per liter (umol/L)
Change in serum uric acid | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (umol/L)
Change in total bilirubin | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (umol/L)
Change in alanine aminotransferase (ALT) | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline in international units per liter (IU/L)
Change in aspartate transaminase (AST) | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (IU/L)
Change in gamma-glutamyl transpeptidase (GGT) | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (IU/L)
Change in alkaline phosphatase (ALP) | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (IU/L)
Change in serum total protein | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline in grams per liter (g/L)
Change in serum albumin | Measured at weeks 0,4,8,12,13 and follow up (week 14)
  Change from baseline (g/L)
Change in hematocrit | Measured at weeks 0,4,8,12,13 and follow-up (week 14)
  Change from baseline (%)
Change in hemoglobin | Measured at weeks 0,4,8,12,13 and follow-up (week 14)
  Change from baseline (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Heshmati, MD, Study Director — Gelesis, Inc.
Locations (5):
- Czechia (2):
  - Hradec Králové, Hradec
  - Charles University, Prague
- University of Cophenhagen, Copenhagen, Denmark
- Italy (2):
  - Federico University Hospital, Naples
  - Policlinico Umberto I, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Greenway FL, Aronne LJ, Raben A, Astrup A, Apovian CM, Hill JO, Kaplan LM, Fujioka K, Matejkova E, Svacina S, Luzi L, Gnessi L, Navas-Carretero S, Alfredo Martinez J, Still CD, Sannino A, Saponaro C, Demitri C, Urban LE, Leider H, Chiquette E, Ron ES, Zohar Y, Heshmati HM. A Randomized, Double-Blind, Placebo-Controlled Study of Gelesis100: A Novel Nonsystemic Oral Hydrogel for Weight Loss. Obesity (Silver Spring). 2019 Feb;27(2):205-216. doi: 10.1002/oby.22347. Epub 2018 Nov 13. PMID 30421844